CLINICAL TRIAL: NCT04475419
Title: Restoration Quality in Molars Affected by Molar-incisor-hypomineralization Using Composite Restorations or Preformed Metal Crowns: Two-arm Randomized Controlled Trial.
Brief Title: Restoration Quality in Molars Affected by Molar Incisor Hypo Mineralization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud mohamed hassan, Assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01008322329
Record Dates: First submitted 2019-07-31; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: parallel groups
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct composite restorations (Active Comparator): bulk-fill composite (Filtek BulkFlow, 3M Espe) will be used and covered using a nanohybrid composite, (Filtek XT, 3M Espe)
  Interventions: Procedure: preformed stainless steel crowns cemented by glass ionomer luting cement(Ketac Cem, 3M Espe)
- preformed metal crowns (Active Comparator): preformed stainless steel crowns cemented by glass ionomer luting cement(Ketac Cem, 3M Espe)
  Interventions: Procedure: preformed stainless steel crowns cemented by glass ionomer luting cement(Ketac Cem, 3M Espe)

INTERVENTIONS:
Procedure: preformed stainless steel crowns cemented by glass ionomer luting cement(Ketac Cem, 3M Espe) — covering the affected molar with preformed metal crown cemented by glass ionomer luting cement(Ketac Cem, 3M Espe)

SUMMARY:
Restoration quality of molars affected by MIH using two different types of restorations direct composite and preformed crowns

DETAILED DESCRIPTION:
MIH or molar incisor hypomineralization is one of the difficult clinical situations to be managed by dentists the aim of this study is to specify which is the better treatment among composite restorations and preformed crowns in terms of gingival health patient satisfaction pain hypersensetivity acceptability by the patienat hypersensetivity and the need for future retreatment

ELIGIBILITY:
Inclusion Criteria:

.Children with molar incisor hypo mineralization in one fully erupted molar or more.

* Age ranging from 7-12 years.
* Cooperative children
* Good general health

Exclusion Criteria:

* Patients participating in other experiments .Patients with parents planning to move away within the following year.
* Patients with only mildly affected MIH molars that do not require extensive restorative treatment.
* MIH-affected molars that have a very poor prognosis and require extraction.
* First permanent molars that are affected with other developmental defects, such as hypoplasia, dental fluorosis or amelogenesis imperfecta.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
pain after the restoration .Binary (yes or No) | 12 MONTHS
  questionnaire

SECONDARY OUTCOMES:
Acceptability of the treatment Binary (yes or No) | 12 months
  questionnaire
restoration quality Score index | 12 months
  (FDI criteria; criterion marginal adaptation)
health-related quality of life changes by the therapies | 12 months
  measured as difference in Child Perceptions Questionnaire CPQ 8-10/11-14)

CONTACTS AND LOCATIONS:
Overall Officials: manalf M elshiekh, MASTER, Study Chair — CU

IPD SHARING:
Plan to Share IPD: No